CLINICAL TRIAL: NCT06051006
Title: The Value of Electrical Stapedial Reflex Thresholds (eSRTs) in Determining Upper Stimulation Levels in Cochlear Implant Maps
Brief Title: The Value Electrical Stapedial Reflex Thresholds (eSRTs) Cochlear Implant Mapping
Acronym: eSRT
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230584; 2023-A00644-41 (Other: IDRCB Number)
Record Dates: First submitted 2023-07-18; First posted 2023-09-22 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Profound Hearing Loss; Cochlear Implants
Keywords: Profound hearing loss; Cochlear implants; Cochlear implant programming; Stapedial reflex

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Minor patients from 8 years with cochlear implants for at least 1 year and followed at Hôpital Necker-Enfants malades.
  Interventions: Other: ESR and ECAP measurements; Other: Device setting; Other: Speech audiometry; Other: Intelligibility in noise test; Other: Cochlear implant datalogging, speech audiometry test, FraSimat test

INTERVENTIONS:
Other: ESR and ECAP measurements — Measurement of electrically evoked stapedial reflexes (ESRT) by stimulation via the cochlear implant. Measurement of the Electric compound action potentials (ECAPs) on the electrodes where the ESRT were performed.
  The measurements and tests will be performed during a routine visit to the Necker hospital for the adjustment of the cochlear implant (visit 1).
Other: Device setting — The adjustment will be made by an audioprosthetist at the Center for Research in Audiology at Necker Hospital. The purpose of this setting is to modify the comfort thresholds using the ESR via a correction (according to the literature). The cochlear implant (CI) will therefore be set with the setting using the ESR (setting 2). The basic setting (setting 1) will be stored in memory in the CI. If ever the patient does not support setting 2, he/she will have the possibility of returning to the basic setting, without having to return to the Necker hospital for an additional setting.
  The measurements and tests will be done during an usual visit of the patient to the Necker hospital for the adjustment of the cochlear implant (visit 1).
Other: Speech audiometry — This examination is part of the usual care for a patient with a cochlear implant. Fournier's monosyllabic test will be used. The test will be carried out by an audioprosthetist at the Center for Research in Audiology at Necker Hospital. The measurement will be performed under both setting conditions: setting 1 (current setting) and setting 2 (based on ESR). The order of administration will be randomized in order to overcome a training effect.
  The measurements and tests will be done during an usual visit of the patient to the Necker hospital for the adjustment of the cochlear implant (visit 1).
Other: Intelligibility in noise test — The FraSimat is a measure of speech perception in noise. The test consists of 14 sentences of 3 words, recorded in the presence of background noise, which the child must listen to and repeat. The background noise remains fixed at 65dB HL and the speech intensity adapts according to the patient's responses. The measurement will be performed under two setting conditions: MAP 1 (current setting) and MAP 2 (setting based on ESR). The order of administration will be randomized in order to overcome a training effect.
  The measurements and tests will be done during an usual visit of the patient to the Necker hospital for the adjustment of the cochlear implant (visit 1).
  Other Names: FraSimat
Other: Cochlear implant datalogging, speech audiometry test, FraSimat test — The follow-up visit (visit 2) will take place 1 month after visit 1 only for patients with a comfort levels threshold (via the eSRT) different from the current threshold (C-subjective).
  At the start of the visit, cochlear implant datalogging will be recorded to determine the use of both settings (setting 2, using the ESR and setting 1, basic setting) while wearing the cochlear implant.
  The datalogging will be recorded by an audioprosthetist at the Center for Research in Audiology at Necker Hospital.
  If the patient has worn the new program (setting 2), the speech audiometry test and the FraSimat test (Intelligibility in noise test) will be performed again with the setting based on ESR.

SUMMARY:
One of the most significant challenges in cochlear implant programming, particularly for very young children and those with an associated pathologies, is the measurement of subjective comfort levels (= C-Subjective). Currently, to define this C-Subjective level, patients are presented with a loudness scale and must indicate whether the sound stimulus, sent via the implant, is soft, comfortable, or loud. The lower and upper stimulation levels must be determined for each electrode in order to program the implant. For many patients this can be difficult due to a lack of auditory experience and confusion between the sensation of sound intensity (weak or loud) and frequency (low or high).

A less commonly used but more objective approach to programming upper stimulation levels involves the use of the electrical stapedial reflex threshold (eSRTs) value. eSRTs are a promising measure, given the demonstrated correlation between the threshold that generates a stapedial reflex and the C-subjective level. Furthermore, eSRTs can be recorded in the majority of patients, and can typically be evoked at a comfortable stimulation level i.e. inferior to the uncomfortable level.

The main objective of this study is investigate the link between subjective comfort levels (C-subjective levels) and the eSRT.

DETAILED DESCRIPTION:
One of the most significant challenges in cochlear implant programming, particularly for very young children and those with an associated pathologies, is the measurement of subjective comfort levels (= C-Subjective). Currently, to define this C-Subjective level, patients are presented with a loudness scale and must indicate whether the sound stimulus, sent via the implant, is soft, comfortable, or loud. The lower and upper stimulation levels must be determined for each electrode in order to program the implant. For many patients this can be difficult due to a lack of auditory experience and confusion between the sensation of sound intensity (weak or loud) and frequency (low or high).

For these patients, the adjustment is often based on the dynamic range recommended by the manufacturer in relation to the threshold (lower stimulation level) and/or on the discomfort level (upper stimulation level).

Objective measures such as ECAPs (Electric compound action potentials) are commonly used to estimate upper stimulation levels.

These measurements are useful for confirming electrode function and neuronal response, and some research has shown that these measures are correlated with the upper stimulation level. However, other studies suggest that ECAPs are poor predictors of high (and low) stimulation levels and can show variability between electrodes and between subjects.

A less commonly used but more objective approach to programming upper stimulation levels involves the use of the electrical stapedial reflex threshold (eSRTs) value. eSRTs are a promising measure, given the demonstrated correlation between the threshold that generates a stapedial reflex and the C-subjective level. Furthermore, eSRTs can be recorded in the majority of patients, and can typically be evoked at a comfortable stimulation level i.e. inferior to the uncomfortable level.

The patient settings are known as the MAP, where the upper and lower levels of stimulation are defined.

MAPs using eSRTs to set upper stimulation levels (C-eSRT) have been shown equal or better speech recognition results compared to behavior-based MAPs (intensity scale). Additionally, eSRT-based MAPs have been shown to result in equal sound intensity across all electrodes, and patients tend to prefer eSRT-based MAPs over behavioral MAPs.

The main objective of this study is investigate there is a link between subjective comfort levels (C-subjective levels) and the eSRT.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 8-17 years at the time of inclusion with cochlear implants for at least 1 year and followed at Hôpital Necker-Enfants malades
* Use oral French as the main mode of communication
* Have a tonal threshold with the cochlear implant of 40 dB or more
* Have a normal tympanogram
* Have a voice threshold of less than 70% at 30dB HL
* Information and non-opposition of holders of parental authority and minor patients to participate in the study

Exclusion Criteria:

* Present a severe neurological pathology before inclusion (which can be identified by an MRI +/- a neuro-pediatric assessment)
* Present, on inclusion, a cognitive or psychiatric impairment or severe developmental delay
* Be part of a family that does not understand oral French
* Patients under AME (State Medical Aid)

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Minor patients from 8 years with cochlear implants for at least 1 year and followed by a physician at Hôpital Necker-Enfants malades.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2026-01-07 (Estimated); Study Completion 2026-01-07 (Estimated)

PRIMARY OUTCOMES:
The relationship between the patient's current upper stimulation level (C-subjective) and the measured eSRT | Day 0
  Correlation between the patient's current upper stimulation level (C-subjective) and the measured eSRT measured at the visit 1.

SECONDARY OUTCOMES:
To determine the relationship between the difference between C-subjective and the eSRT and the speech recognition scores | Day 0
  Correlation between the difference between C-subjective and the eSRT measured at the visit 1 and the percent correct on the Fournier's monosyllabic word test.
To determine the relationship between the ECAPs (electric compound action potentials) and the eSRT | Day 0
  Correlation between the patient's ECAPs (electric compound action potentials) and the measured eSRT measured at the visit 1.
To evaluate the difference in speech performance in silence obtained using a C-subjective MAP and a C-eSRT MAP | 1 month
  Comparison of the percent correct on the Fournier's monosyllabic word test at the visit 1, using the C-subjective MAP and at the visit 2, using the C-eSRT MAP.
To evaluate the difference in speech performance in noise obtained using a C-subjective MAP and a C-eSRT MAP | 1 month
  Comparison of the percent correct on the FraSimat speech in noise test at the visit 1, using the C-subjective MAP and at the visit 2, using the C-eSRT MAP.
The difference in average daily use time of C-subjective MAP and a C-eSRT MAP | 1 month
  Comparison of the number of average daily hours of use time for the C-subjective MAP and the C-eSRT MAP at the visit 2.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa MacAskill, Study Director — Assistance Publique - Hôpitaux de Paris; Nara Vaez-Leppin, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allum JH, Greisiger R, Probst R. Relationship of intraoperative electrically evoked stapedius reflex thresholds to maximum comfortable loudness levels of children with cochlear implants. Int J Audiol. 2002 Mar;41(2):93-9. doi: 10.3109/14992020209090399. PMID 12212861
- [Background] Walkowiak A, Lorens A, Polak M, Kostek B, Skarzynski H, Szkielkowska A, Skarzynski PH. Evoked stapedius reflex and compound action potential thresholds versus most comfortable loudness level: assessment of their relation for charge-based fitting strategies in implant users. ORL J Otorhinolaryngol Relat Spec. 2011;73(4):189-95. doi: 10.1159/000326892. Epub 2011 Jun 10. PMID 21659787
- [Background] Geers A, Brenner C, Davidson L. Factors associated with development of speech perception skills in children implanted by age five. Ear Hear. 2003 Feb;24(1 Suppl):24S-35S. doi: 10.1097/01.AUD.0000051687.99218.0F. PMID 12612478
- [Background] Brown CJ, Abbas PJ, Gantz B. Electrically evoked whole-nerve action potentials: data from human cochlear implant users. J Acoust Soc Am. 1990 Sep;88(3):1385-91. doi: 10.1121/1.399716. PMID 2229673
- [Background] Brown CJ, Hughes ML, Luk B, Abbas PJ, Wolaver A, Gervais J. The relationship between EAP and EABR thresholds and levels used to program the nucleus 24 speech processor: data from adults. Ear Hear. 2000 Apr;21(2):151-63. doi: 10.1097/00003446-200004000-00009. PMID 10777022
- [Background] Gordon KA, Papsin BC, Harrison RV. Toward a battery of behavioral and objective measures to achieve optimal cochlear implant stimulation levels in children. Ear Hear. 2004 Oct;25(5):447-63. doi: 10.1097/01.aud.0000146178.84065.b3. PMID 15599192
- [Background] Hodges AV, Butts S, Dolan-Ash S, Balkany TJ. Using electrically evoked auditory reflex thresholds to fit the CLARION cochlear implant. Ann Otol Rhinol Laryngol Suppl. 1999 Apr;177:64-8. doi: 10.1177/00034894991080s413. PMID 10214804
- [Background] Hodges AV, Balkany TJ, Ruth RA, Lambert PR, Dolan-Ash S, Schloffman JJ. Electrical middle ear muscle reflex: use in cochlear implant programming. Otolaryngol Head Neck Surg. 1997 Sep;117(3 Pt 1):255-61. doi: 10.1016/s0194-5998(97)70183-9. PMID 9334774
- [Background] Lorens A, Walkowiak A, Piotrowska A, Skarzynski H, Anderson I. ESRT and MCL correlations in experienced paediatric cochlear implant users. Cochlear Implants Int. 2004 Mar;5(1):28-37. doi: 10.1002/cii.121. PMID 18792192
- [Background] Van Den Abbeele T, Noel-Petroff N, Akin I, Caner G, Olgun L, Guiraud J, Truy E, Attias J, Raveh E, Belgin E, Sennaroglu G, Basta D, Ernst A, Martini A, Rosignoli M, Levi H, Elidan J, Benghalem A, Amstutz-Montadert I, Lerosey Y, De Vel E, Dhooge I, Hildesheimer M, Kronenberg J, Arnold L. Multicentre investigation on electrically evoked compound action potential and stapedius reflex: how do these objective measures relate to implant programming parameters? Cochlear Implants Int. 2012 Feb;13(1):26-34. doi: 10.1179/1754762810Y.0000000001. PMID 22340749
- [Background] Brickley G, Boyd P, Wyllie F, O'Driscoll M, Webster D, Nopp P. Investigations into electrically evoked stapedius reflex measures and subjective loudness percepts in the MED-EL COMBI 40+ cochlear implant. Cochlear Implants Int. 2005 Mar;6(1):31-42. doi: 10.1002/cii.18. PMID 18792318
- [Background] Craddock L, Cooper H, van de Heyning P, Vermeire K, Davies M, Patel J, Cullington H, Ricaud R, Brunelli T, Knight M, Plant K, Dees DC, Murray B. Comparison between NRT-based MAPs and behaviourally measured MAPs at different stimulation rates--a multicentre investigation. Cochlear Implants Int. 2003 Dec;4(4):161-70. doi: 10.1179/cim.2003.4.4.161. PMID 18792149
- [Background] Franck KH, Norton SJ. Estimation of psychophysical levels using the electrically evoked compound action potential measured with the neural response telemetry capabilities of Cochlear Corporation's CI24M device. Ear Hear. 2001 Aug;22(4):289-99. doi: 10.1097/00003446-200108000-00004. PMID 11527036
- [Background] Jeon EK, Brown CJ, Etler CP, O'Brien S, Chiou LK, Abbas PJ. Comparison of electrically evoked compound action potential thresholds and loudness estimates for the stimuli used to program the Advanced Bionics cochlear implant. J Am Acad Audiol. 2010 Jan;21(1):16-27. doi: 10.3766/jaaa.21.1.3. PMID 20085196
- [Background] Joly CA, Pean V, Hermann R, Seldran F, Thai-Van H, Truy E. Using Electrically-evoked Compound Action Potentials to Estimate Perceptive Levels in Experienced Adult Cochlear Implant Users. Otol Neurotol. 2017 Oct;38(9):1278-1289. doi: 10.1097/MAO.0000000000001548. PMID 28834942
- [Background] Smoorenburg GF, Willeboer C, van Dijk JE. Speech perception in nucleus CI24M cochlear implant users with processor settings based on electrically evoked compound action potential thresholds. Audiol Neurootol. 2002 Nov-Dec;7(6):335-47. doi: 10.1159/000066154. PMID 12401965
- [Background] Wolfe J, Kasulis H. Relationships among objective measures and speech perception in adult users of the HiResolution Bionic Ear. Cochlear Implants Int. 2008 Jun;9(2):70-81. doi: 10.1179/cim.2008.9.2.70. PMID 18680210
- [Background] Bresnihan M, Norman G, Scott F, Viani L. Measurement of comfort levels by means of electrical stapedial reflex in children. Arch Otolaryngol Head Neck Surg. 2001 Aug;127(8):963-6. doi: 10.1001/archotol.127.8.963. PMID 11493206
- [Background] Polak M, Hodges AV, King JE, Payne SL, Balkany TJ. Objective methods in postlingually and prelingually deafened adults for programming cochlear implants: ESR and NRT. Cochlear Implants Int. 2006 Sep;7(3):125-41. doi: 10.1179/cim.2006.7.3.125. PMID 18792380
- [Background] Holder JT, Holcomb MA, Snapp H, Labadie RF, Vroegop J, Rocca C, Elgandy MS, Dunn C, Gifford RH. Guidelines for Best Practice in the Audiological Management of Adults Using Bimodal Hearing Configurations. Otol Neurotol Open. 2022 Jun;2(2):e011. doi: 10.1097/ONO.0000000000000011. Epub 2022 Jun 24. PMID 36274668
- [Background] Palani S, Alexander A, Sreenivasan A. Evaluation of the Electrically-Evoked Stapedial Reflex Threshold in Pediatric Cochlear Implant Users with High-Frequency Probe Tones. Int Arch Otorhinolaryngol. 2022 Feb 8;26(4):e566-e573. doi: 10.1055/s-0042-1742332. eCollection 2022 Oct. PMID 36405469